CLINICAL TRIAL: NCT00348946
Title: Androgen Effect on Motor/Cognitive Outcome in Klinefelter Syndrome
Brief Title: Androgen Effect on Klinefelter Syndrome Motor Outcome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01NS050597-01A2 (NIH)
Record Dates: First submitted 2006-07-03; First posted 2006-07-06 (Estimated); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Klinefelter Syndrome
Keywords: Klinefelter syndrome; androgen; androgen oxandrolone
MeSH Terms: conditions — Klinefelter Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxandrolone (Active Comparator): Androgen oxandrolone: Oxandrolone, 0.6 > mg/kg/day, orally, for 2 years.
  Interventions: Drug: androgen oxandrolone
- Placebo (Placebo Comparator): An inactive substance.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: androgen oxandrolone — Oxandrolone ,06 >mg/kg/day, orally, for 2 years
  Arms: Oxandrolone
Other: placebo — an inactive substance
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of low-dose androgen on the motor and cognitive development of boys with Klinefelter syndrome.

DETAILED DESCRIPTION:
Klinefelter syndrome (KS), a genetic disorder that affects males only, is characterized by having an extra X chromosome. The phenotype - or physical and learning features - includes testicular failure, tall stature, and specific cognitive and behavioral attributes such as diminished motor function, language-based learning difficulties, poor self-image, and shyness. The KS phenotype may be the result of androgen deficiency in utero, infancy, and childhood. For individuals with KS, androgen replacement is standard treatment in adolescence and adulthood but has not been used earlier in childhood or included in the standard medical care of KS children ages 4 to 12.

The purpose of this study is to examine the effects of androgen on learning and development in boys with KS. Researchers also want to determine if low-dose androgen replacement at an early age will improve some of the learning difficulties associated with the disorder. The overall goal of this study is to address questions regarding the relationship of early androgen deficiency to learning and motor function.

Participants in the study will be randomized to one of two treatment groups, receiving either oxandrolone (low-dose androgen) or placebo, for two years. All participants will be evaluated for safety at the beginning of the study and at 3, 6, 12, 18, and 24 months. Also at the beginning of the study and every 3 to 6 months thereafter (for a total of 6 visits), the researchers will perform a careful history and physical examination and a bone age X-ray, and obtain a blood sample.

Participation in the trial will last two years and includes 6 clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Karyotype diagnosis of Klinefelter syndrome
* Chronological age of 4-12 years
* No treatment with androgen in the past year

Exclusion Criteria:

* Major liver, kidney or other systemic disease
* Variant karyotypes including 47,XYY males
* Evidence of spontaneous onset of puberty, defined as testicular size > 4ml

Ages: 4 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2006-07; Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith L. Ross, M.D., Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Department of Pediatrics, 1025 Walnut Street, Suite 726, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Davis SM, Lahlou N, Cox-Martin M, Kowal K, Zeitler PS, Ross JL. Oxandrolone Treatment Results in an Increased Risk of Gonadarche in Prepubertal Boys With Klinefelter Syndrome. J Clin Endocrinol Metab. 2018 Sep 1;103(9):3449-3455. doi: 10.1210/jc.2018-00682. PMID 29931143
- [Derived] Ross JL, Kushner H, Kowal K, Bardsley M, Davis S, Reiss AL, Tartaglia N, Roeltgen D. Androgen Treatment Effects on Motor Function, Cognition, and Behavior in Boys with Klinefelter Syndrome. J Pediatr. 2017 Jun;185:193-199.e4. doi: 10.1016/j.jpeds.2017.02.036. Epub 2017 Mar 10. PMID 28285751
- [Derived] Davis S, Lahlou N, Bardsley M, Temple MC, Kowal K, Pyle L, Zeitler P, Ross J. Gonadal function is associated with cardiometabolic health in pre-pubertal boys with Klinefelter syndrome. Andrology. 2016 Nov;4(6):1169-1177. doi: 10.1111/andr.12275. Epub 2016 Sep 16. PMID 27637014

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxandrolone: androgen oxandrolone: Oxandrolone ,0.6 >mg/kg/day, orally, for 2 years.
Period: Overall Study
Arm/Group | Oxandrolone | Placebo
Started | 46 | 47
Completed | 35 | 35
Not Completed | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxandrolone | Placebo | Total
Number analyzed (Participants) | 46 | 47 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 46 | 47 | 93
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.9 (2.2) | 8.5 (2.6) | 7.7 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 46 | 47 | 93
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 33 | 34 | 67
  Ethnicity: African American | 6 | 6 | 12
  Ethnicity: Hispanic | 5 | 3 | 8
  Ethnicity: Asian/Pacific Islander | 2 | 3 | 5
  Ethnicity: Other | 0 | 1 | 1
Tanner 1 pubic hair [Count of Participants; unit: Participants] | 43 | 38 | 81
BMI Standard Deviation Score (SDS) [Mean (Standard Deviation); unit: kg/m^2] | 0.40 (1.15) | 0.58 (1.17) | 0.49 (1.16)
Waist circumference percentile >75 percentile [Count of Participants; unit: Participants] | 17 | 22 | 39
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] | 167 (33) | 162 (27) | 164 (29)
LDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 106 (31) | 104 (24) | 104.4 (25.4)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 75.4 (58.2) | 67.7 (32.6) | 70.7 (46)
Triglycerides > 100 mg/dL [Count of Participants; unit: Participants] | 9 | 6 | 15
HDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 46 (10.4) | 44.8 (10.1) | 45.7 (10)
HDL cholesterol < 50 mg/dL [Count of Participants; unit: Participants] | 31 | 31 | 62
Fasting blood glucose, mg/dL [Mean (Standard Deviation); unit: mg/dL] | 84.8 (8.4) | 85.2 (6.7) | 85.2 (7.6)
Fasting blood glucose > 110 mg/dL [Count of Participants; unit: Participants] | 1 | 0 | 1
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 87.2 (9.7) | 90.9 (9.4) | 88.7 (9.6)
Systolic blood pressure > 90th percentile for age and height [Count of Participants; unit: Participants] | 0 | 0 | 0
Diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 52.3 (6.9) | 56.9 (7.3) | 55 (8.5)
Diastolic blood pressure > 90th percentile for age and height [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Motor Function/Strength
Description: Outcome measures were tested using the following assessments: Bruininks-Osertesky Test of Motor Proficiency (BOT) subscales of (1) Visual Motor Control, (2) Upper limb Speed, and (3) Strength, Physical and Neurological Evaluation for Soft Signs (PANESS), and Hand Strength Dynamometer. BOT assess the child's motor development and includes standard scores (mean=100, SD=15) and subtest scores and is normed for sex and age (4-14.5 years). PANESS assesses the time required to press thumb to 4 fingers 20 times for the dominant and nondominant hands and includes standard scores (mean=100, SD=15) with age-specific norms (4-18 years). Hand strength dynamometer assess hand strength in the dominant and nondominant hands and includes standard scores (mean=100, SD=15). Data is expressed as standard scores with mean of 100 and SD of 15. The minimum standard score is 50; the maximum standard score is 145. Higher scorers imply better function.
Time Frame: 2 years per subject
Population: Some participants were not able to complete all test and/or it was determined by the investigator that their results do reflect their ability and they were removed from the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxandrolone | Placebo
Number analyzed (Participants) | 35 | 36
score on a scale
  BOT Visual-motor control SS | 86 (1) | 81 (1)
  BOT Upper limb speed SS | 92 (1) | 89 (2)
  BOT Strength SS | 88 (1) | 85 (1)
  Hand Dynamometer SS- dominant hand: number analyzed (Participants) | 34 | 36
  Hand Dynamometer SS- dominant hand | 123 (2) | 118 (2)
  PANESS SS- dominant hand: number analyzed (Participants) | 21 | 24
  PANESS SS- dominant hand | 91 (3) | 91 (3)
Statistical Analysis 1: Comparison: Oxandrolone vs Placebo; Test type: Superiority — BOT Visual-motor control; p = 0.005, ANCOVA
Statistical Analysis 2: Comparison: Oxandrolone vs Placebo; BOT upper limb speed; Test type: Superiority; p = 0.17, ANCOVA
Statistical Analysis 3: Comparison: Oxandrolone vs Placebo; BOT strength; Test type: Superiority; p = 0.17, ANCOVA
Statistical Analysis 4: Comparison: Oxandrolone vs Placebo; Hand dynamometer; Test type: Superiority; p = 0.06, ANCOVA
Statistical Analysis 5: Comparison: Oxandrolone vs Placebo; PANESS; Test type: Superiority; p = 0.87, ANCOVA

2. Secondary Outcome: Cognitive Function and Language
Description: Outcome measures were tested using the Differential Ability Scales - 2nd edition (DAS-II). DAS-II provides an age- and sex-standardized assessment of intellectual functioning (General Concept Ability subscale similar to IQ) in children ages 2-17 years of age (mean=100, SD=15). The Verbal Cluster measures the child's ability to define words and perform verbal reasoning tasks. The Nonverbal Cluster measures the child's inductive and sequential reasoning abilities. The Spatial Cluster measures visuospatial construction ability, spatial memory, and spatial reasoning. Data is expressed as standard scores with mean of 100 and SD of 15. The minimum standard score is 50; the maximum standard score is 145. Higher scores imply better function.
Time Frame: 2 years per subject
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxandrolone | Placebo
Number analyzed (Participants) | 35 | 36
score on a scale
  DAS: General Concept Ability | 96 (2) | 94 (2)
  DAS: Verbal Cluster | 92 (2) | 90 (2)
  DAS: Nonverbal Cluster | 102 (2) | 101 (2)
  DAS: Spatial Cluster | 96 (2) | 94 (2)
Statistical Analysis 1: Comparison: Oxandrolone vs Placebo; DAS: General concept ability; Test type: Superiority; p = 0.44, ANCOVA
Statistical Analysis 2: Comparison: Oxandrolone vs Placebo; DAS: Verbal Cluster; Test type: Superiority; p = 0.57, ANCOVA
Statistical Analysis 3: Comparison: Oxandrolone vs Placebo; DAS: Nonverbal Cluster; Test type: Superiority; p = 0.55, ANCOVA
Statistical Analysis 4: Comparison: Oxandrolone vs Placebo; DAS: Spatial Cluster; Test type: Superiority; p = 0.65, ANCOVA

3. Secondary Outcome: Working Memory/Attention
Description: Outcome measures were tested using the following cognitive assessments: Digit Span Backward, A Neuropsychological Assessment (NEPSY) subscales of (1) Phonemic Fluency and (2) Semantic Fluency, and Connors' Continuous Performance Test (CPT-II) subscales (1) Omissions, (2) Commissions, (3) Hit Reaction, (4) Variability, and (5) Preservations. Digit Span Backward tests working memory and is normed for children ages 5-16 years. Phonemic Fluency measures the number of words that the child can name beginning with the letters F and S (ages 6-12). Semantic Fluency measures the number of words the child can name in the categories food and drink (ages 4-12). CPT-II measures the ability to maintain attention over an extended period of time. All scores are reported as standard scores with a mean of 100 and SD of 15. The minimum standard score is 50; the maximum standard score is 145. Higher scores imply better function.
Time Frame: 2 years per participant
Population: Some participants were not able to complete all assessments and/or it was determined by the investigator that their results do reflect their ability and they were removed from the analysis .
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxandrolone | Placebo
Number analyzed (Participants) | 32 | 33
score on a scale
  Digit span backward: number analyzed (Participants) | 29 | 33
  Digit span backward | 96 (2) | 92 (2)
  Phonemic fluency: number analyzed (Participants) | 12 | 17
  Phonemic fluency | 95 (3) | 91 (2)
  Semantic fluency: number analyzed (Participants) | 12 | 17
  Semantic fluency | 99 (4) | 94 (3)
  CPT: omissions: number analyzed (Participants) | 32 | 31
  CPT: omissions | 88 (4) | 83 (4)
  CPT: commissions: number analyzed (Participants) | 32 | 31
  CPT: commissions | 101 (2) | 100 (2)
  CPT: hit reaction time: number analyzed (Participants) | 32 | 31
  CPT: hit reaction time | 84 (3) | 80 (3)
  CPT variability: number analyzed (Participants) | 32 | 31
  CPT variability | 86 (2) | 86 (2)
  CPT: preservations: number analyzed (Participants) | 32 | 31
  CPT: preservations | 76 (5) | 74 (5)
Statistical Analysis 1: Comparison: Oxandrolone vs Placebo; Digit Span backward; Test type: Superiority; p = 0.23, ANCOVA
Statistical Analysis 2: Comparison: Oxandrolone vs Placebo; Phonetic fluency; Test type: Superiority; p = 0.36, ANCOVA
Statistical Analysis 3: Comparison: Oxandrolone vs Placebo; Semantic fluency; Test type: Superiority; p = 0.37, ANCOVA
Statistical Analysis 4: Comparison: Oxandrolone vs Placebo; CPT: omissions; Test type: Superiority; p = 0.41, ANCOVA
Statistical Analysis 5: Comparison: Oxandrolone vs Placebo; CPT: commissions; Test type: Superiority; p = 0.73, ANCOVA
Statistical Analysis 6: Comparison: Oxandrolone vs Placebo; CPT: hit reaction time; Test type: Superiority; p = 0.40, ANCOVA
Statistical Analysis 7: Comparison: Oxandrolone vs Placebo; CPT: variability; Test type: Superiority; p = 0.95, ANCOVA
Statistical Analysis 8: Comparison: Oxandrolone vs Placebo; CPT: preservations; Test type: Superiority; p = 0.78, ANCOVA

4. Secondary Outcome: Psychosocial and Behavior Domain
Description: Outcome measures were tested using the following social assessments: The Child Behavior Checklist (CBCL) and The Children's Depression Inventory (CDI). The CBCL is standardized measure of behavior problems and social competency normed for children ages 4-16. Higher scores indicate more problems, with the cutoff for the clinical range at a t score greater than or equal to 67. The CDI assess cognitive, affective and behavioral signs of depression in children ages 6-17. The CDI total score reflects the presence of overall depressive symptoms. All scores are expressed as t-scores with a mean of 50 and SD of 10. Lower scores imply better function and higher scores indicate more problem behaviors.
Time Frame: 2 years per participants
Population: Some participants were not able to complete all assessments and/or it was determined by the investigator that their results do reflect their ability and they were removed from the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxandrolone | Placebo
Number analyzed (Participants) | 35 | 36
score on a scale
  CBCL: behavior total t-score | 56 (1) | 59 (1)
  CBCL: internalizing total t-score | 54 (1) | 57 (1)
  CBCL: externalizing total t-score | 51 (2) | 54 (1)
  CDI: total t-score: number analyzed (Participants) | 15 | 21
  CDI: total t-score | 45 (2) | 47 (2)
Statistical Analysis 1: Comparison: Oxandrolone vs Placebo; CBCL: Behavior total; Test type: Superiority; p = 0.16, ANCOVA
Statistical Analysis 2: Comparison: Oxandrolone vs Placebo; CBCL: Internalizing total; Test type: Superiority; p = 0.10, ANCOVA
Statistical Analysis 3: Comparison: Oxandrolone vs Placebo; CBCL: externalizing total; Test type: Superiority; p = 0.24, ANCOVA
Statistical Analysis 4: Comparison: Oxandrolone vs Placebo; CDI: Total; Test type: Superiority; p = 0.50, ANCOVA

5. Secondary Outcome: Psychosocial and Behavior Domain
Description: Outcome measures were tested using The Piers-Harris Self Concept Scale. Scoring provides a total standard score and scores on six subscales: physical appearance and attributes, freedom from anxiety, intellectual and school status, behavioral adjustment, happiness and satisfaction, and popularity. Subscales are summed and standardized to provide the total standard score with a mean of 100 and SD of 15. The minimum standard score is 50; the maximum standard score is 145. Higher scores imply better function.
Time Frame: 2 years per subject
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxandrolone | Placebo
Number analyzed (Participants) | 16 | 20
units on a scale | 105 (3) | 100 (2)
Statistical Analysis 1: Comparison: Oxandrolone vs Placebo; Test type: Superiority; p = 0.15, ANCOVA

ADVERSE EVENTS:
Time Frame: Two years
Arm/Group | Oxandrolone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/47
Other Adverse Events (participants affected / at risk) | 36/46 | 38/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxandrolone (N=46) | Placebo (N=47)
Musculoskeletal complaints (Musculoskeletal and connective tissue disorders) | 29 (54) | 29 (53)
Infections (any) (Infections and infestations) | 36 (77) | 38 (77)
Headache (Nervous system disorders) | 21 (56) | 22 (42)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Emergency room visits - Musculoskeletal (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Emergency room visits - Asthma/allergy (Immune system disorders) | 3 (4) | 0 (0)
Emergency room visits - Gastrointestinal (Gastrointestinal disorders) | 2 (2) | 1 (1)
Emergency room visits (Nervous system disorders) | 2 (2) | 1 (1)
Emergency room visits (Infections and infestations) | 3 (4) | 3 (3)
Emergency room visits - other (General disorders) | 1 (1) | 1 (1)
Hospitalizations - Medical (General disorders) | 1 (1) | 1 (1)
Hospitalizations - Psychiatric (Psychiatric disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-01-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT00348946/Prot_SAP_000.pdf